CLINICAL TRIAL: NCT03213379
Title: Assessment of Actigraphy Procedures on the Initiation of an Apomorphine Treatment Delivered Through a Pump to Patients With Parkinson's Disease
Acronym: @ctipark
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Orkyn' (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P1530; Ref ID-RCB (Other: 2016-A00261-50)
Record Dates: First submitted 2017-06-15; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Parkinson Disease
Keywords: actimeter; apomorphin pump
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: A unique code is given to each patient enrolled in the study. Neither the name nor the surname of patient are mentioned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Referent group (No Intervention): The patient of the referent group will have 2 measures of actimetry:
  A first one at baseline before the apomorphim set-up:the report will be provided to the investigator and a second one before the 6 months follow-up visit but this report will not be provided to the investigator.
- Actimetry group (Experimental): The patient of the Actimetry group will have at least 4 measures of actimetry and the reports will be all provided to the investigator:
  One at baseline before the apomorphim set-up/ the second one 8 days after the hospitalisation/ the third one 28 days after the hospitalisation and the last one before the 6 months follow-up visit One optional measure can be performed 84 days after the hospitalisation.
  Interventions: Device: Actimetry measures

INTERVENTIONS:
Device: Actimetry measures — The patient will wear actigraphy bracelet during a week that will enable to record patients' movements. The report based on the recording will provide an assessment of daytime somnolence and an indication of propensity for impulsive behaviours.The intervention consisted in 2 supplementary actimetry measures and sending of the actimetry reports to the investigator.
  Arms: Actimetry group

SUMMARY:
The goal of the study is to compare the impact of different actigraphy procedures on the healthcare organization of Parkinson's disease (PK) patients using an apomorphine pump. To do so, the study design includes a patients' randomisation in two groups that will be followed during 6 months.

DETAILED DESCRIPTION:
The two groups are:

Referent group with one actimetric report at baseline Actimetry group with one actimetric report at baseline and during the follow-up. Using these reports the investigator will be able to modify the prescription of the apomorphin pump without seeing the patient.

It is planned to follow the patients during 6 months of follow-up and 3 medical visits will be conducted as per the standard practice:

1 visit before the installation of the pump

1 visit after the pump installation straight after the patient comes out the hospital

1 visit at 6 months

ELIGIBILITY:
Inclusion Criteria:

Adult suffering from Parkinson's disease aged up to 75 years (included) Patient for whom a first set-up of an apomorphine pump has been decided under medical guidelines Patient who chose the OPTIPARK package (ORKYN nurses) Patient willing to wear the actigraphy bracelet as per the protocol Patient who read, understood and signed the consent form.

Exclusion Criteria:

Patient not willing to take part in the study Patient who had a previous set-up of an apomorphine pump Patient with dementia Dependant patients or patients living in institutional care Patient with a temporary pump of apomorphine compromising a six months follow-up Patient with non-major motor fluctuations Patient already enrolled in an interventional study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-09-15 (Estimated); Study Completion 2018-09-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of the impact of different actigraphy procedures on the healthcare organization of Parkinson's disease (PK) patients using an apomorphine pump | 6 months
  Proportion of patients with an unscheduled healthcare use during the first 6 months of treatment with the pump (after hospitalization for initiation) including: All medical visits to the neurologist due to the Parkinson disease New hospitalization related to the Parkinson disease

IPD SHARING:
Plan to Share IPD: No
There is no plan